CLINICAL TRIAL: NCT05311241
Title: Observational Study of the Use of the Service Giving Access to Teleconsultation in France by Telemedicine Companies
Brief Title: Teleconsultation in Ambulatory Care in France
Acronym: TELET
Status: Completed | Type: Observational
Sponsor: Les Entreprises de Télémédecine (Other)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Telehealth; Telemedicine; Teleconsultation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Teleconsultation is a telemedicine medical act carried out remotely via information and communication technologies. This medical procedure has been legal in France since 2010 and reimbursed by the National Health Insurance under certain conditions since 2018. In 2020, following the COVID-19 epidemic, the lockdowns and the extension of the scope of financial coverage, 17 million teleconsultations have been reimbursed.

To date, few scientific studies have been published in France to precisely describe the use of the service giving access to outpatient teleconsultation, in particular since the major increase in activity linked to the COVID-19 epidemic.

The objective is to describe the use of the service giving access to outpatient teleconsultation carried out in France by teleconsultation companies and compare the use of the teleconsultation service according to the medical density of the territory.

ELIGIBILITY:
Inclusion Criteria:

* Patient who used the teleconsultation access service with one of the telemedicine companies member of the LET participating in the study
* Patient residing in France according to the written information (address and or postal code) given at registration to the telemedicine company
* Teleconsultation service used between August 1, 2021 and November 30, 2021
* Teleconsultation service used in the context of outpatient care (hospitals excluded)
* Teleconsultation service used for a teleconsultation with a doctor registered with the Medical Doctors Council in France

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered with a teleconsultation company member of the LET participating to the study with at least one teleconsultation during the study period.
Sampling Method: Probability Sample
Enrollment: 84000 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Rate of patients without a treating doctor | Through the study completion at the time of the teleconsultation, average 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Julie Salomon, MD, Principal Investigator — Qare
Locations (1):
- Les Entreprises de Télémédecine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohannessian R, Yaghobian S, Simon R, Poinsot-Chaize G, Hiridjee S, Gleize JC, Pierme JP, Amar N, Merlaud C, Maudoux C, Zerah B, Lescure F, Salomon J. Evaluating the Impact of Teleconsultations on Access to Ambulatory Primary Care in Medically Underserved Areas: A National Observational Cross-Sectional Multicenter Study. Telemed J E Health. 2024 Feb;30(2):570-578. doi: 10.1089/tmj.2023.0274. Epub 2023 Aug 29. PMID 37643308